CLINICAL TRIAL: NCT02583126
Title: The Effect and Meaning of a Designed Guided Imagery and Music Intervention on Anticipatory, Acute, and Delayed Side Effect of Chemotherapy in Teenagers With Cancer: a Randomized Controlled Multisite Study
Brief Title: Guided Imagery and Music for the Reduction of Side Effects of Chemotherapy in Teenagers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Danish Cancer Society (Other); Børnecancerfonden (Other); Ronald McDonalds Børnefond (Other); TrygFonden, Denmark (Industry)
Responsible Party: Principal Investigator, Ilan Sanfi, Music therapist, PhD, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GIM-Cancer-Teenagers-1
Record Dates: First submitted 2015-02-03; First posted 2015-10-22 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Cancer
Keywords: Teenager; moderate and/or highly emetogenic chemotherapy
MeSH Terms: conditions — Neoplasms | interventions — Imagery, Psychotherapy; Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Music Group (Experimental): Prescribed medical/chemotherapy treatment plus standard care + Guided Imagery and Music
  Interventions: Behavioral: Guided Imagery and Music
- Control Group (No Intervention): Prescribed medical/chemotherapy treatment plus standard care

INTERVENTIONS:
Behavioral: Guided Imagery and Music — Modified and resource-oriented form of the Bonny Method of Guided Imagery and Music (BM-GIM)
  Other Names: Music and imagery, music therapy, active music listening
  Arms: Music Group

SUMMARY:
The purpose of this study is to determine whether a modified and resource-oriented form of Guided Imagery and Music (GIM) is effective in reducing side effects of chemotherapy in teenagers with cancer.

DETAILED DESCRIPTION:
(Will be added later)

ELIGIBILITY:
Inclusion Criteria:

1. Teenagers at the ages 12-17
2. Four or five (dependent on their overall plan of medical treatment) consecutive courses of chemotherapy administrated at the involved child cancer units and (administered) over a period of minimum 24 hours incl. hydration with assumed moderate to severe nausea and vomiting.

   The specific type of chemotherapy may vary across the four/five consecutive courses but shall include one of the following moderate and/or highly emetogenic types of chemotherapy:

   Moderate emetogenic chemotherapy:
   * Carboplatin
   * Cyclophosphamide <1500 mg/m2
   * Cytarabine >1 g/m2
   * Daunorubicin
   * Doxorubicin
   * Epirubicin
   * Idarubicin
   * Ifosfamide
   * Mitoxantrone
   * Methotrexate >1000 mg/m2

   Highly emetogenic chemotherapy:
   * Cisplatin >25 mg/m2
   * Cyclophosphamide >1500 mg/m2
   * Dacarbazine
3. Understand Norwegian/Danish
4. Read Norwegian/Danish (teenagers or alternatively parents)
5. No significant hearing impairment
6. Informed written consent (teenagers ≥16 years and parents)
7. Subsequent verbal confirmation of written informed consent before enrolment in study

Exclusion Criteria:

1. Previous and/or acute psychiatric diagnosis
2. Cognitive and mental deficits or impaired functioning

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Estimated)
Dates: Start 2014-08; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Duration (minutes) of Acute Nausea | Registered the two first evenings within the first 32 hours after onset of chemotherapy during 5th cycle of chemotherapy after enrolment in study
  Self-reported duration og nausea in minutes during the first 32 hours after onset of chemotherapy

SECONDARY OUTCOMES:
Intensity of Acute Nausea as measured by the Visual Analogue Scale | Registered the two first evenings within the first 32 hours after onset of chemotherapy during 5th cycle of chemotherapy after enrolment in study
  Self-reported intensity of nausea, calculated as the average of the two measurements
Distress regarding Acute Nausea as measured by the Visual Analogue Scale | Registered the two first evenings within the first 32 hours after onset of chemotherapy during 5th cycle of chemotherapy after enrolment in study
  Self-reported distress regarding nausea, calculated as the average of the two measurements
Amount (mg/m2) of Nausea Reducing Medicine Consumed | During admission (an expected average of 3 days) and the first three days after discharge regarding 5th cycle of chemotherapy after enrolment in study
Multiple Acute Side Effects of Chemotherapy as measured by the Memorial Symptom Assessment Scale | Registered the two first evenings within the first 32 hours after onset of chemotherapy during 5th cycle of chemotherapy after enrolment in study
  Self-reported side effects, calculated as the average of the two measurements. The Memorial Symptom Assessment Scale is a self-report composite measure that measures bodily and psychological symptoms of side effects
Numbers of Acute Vomiting | Registered the two first evenings within the first 32 hours after onset of chemotherapy during 5th cycle of chemotherapy after enrolment in study
  Self-reported numbers of vomiting during the first 32 hours
Duration (minutes) of Acute Pain | Registered the two first evenings within the first 32 hours after onset of chemotherapy during 5th cycle of chemotherapy after enrolment in study
  Self-reported duration of acute pain in minutes within the first 32 hours after onset of chemotherapy
Acute Pain Intensity as measured by the Visual Analogue Scale | Registered the two first evenings within the first 32 hours after onset of chemotherapy during 5th cycle of chemotherapy after enrolment in study
  Self-reported intensity of pain, calculated as the average of the two measurements
Number of Days to Absolute Neutrophil Count Recovery defined as ANC ≥ 0.5 x 109/L | Time to Event: Measured Day 1 in 5th cycle of chemotherapy after enrolment in study - until first day with ANC ≥ 0.5 x 109/L after the nadir period (an expected average of 9-15 days)
  Number of days before the immune system recovers after chemotherapy. In the study, Absolute Neutrophil Count Recovery (ANCR) is defined as ANCR ≥ 0.5 x 109/L. In addition, if no nadir < 0.5 x 109/L occurs the period is 0 (zero).
Duration (minutes) of Acute Fatigue | Registered the two first evenings within the first 32 hours after onset of chemotherapy during 5th cycle of chemotherapy after enrolment in study
  Self-reported duration of acute fatigue in minutes within the first 32 hours after onset of chemotherapy
Distress regarding Acute Fatigue as measured by a 5-point Likert-type Scale | Registered the two first evenings within the first 32 hours after onset of chemotherapy during 5th cycle of chemotherapy after enrolment in study
  Self-reported Distress regarding Acute Fatigue, calculated as the average of the two measurements
Appraised food intake and appetite as measured by a 5-point Likert-type Scale | Registered the two first evenings within the first 32 hours after onset of chemotherapy during 5th cycle of chemotherapy after enrolment in study
  Self-reported appraised food intake, calculated as the average of the two measurements
Weight (kg) | Change between weight from during course 1 and course 5 after inclusion in study
Sense of Coherence as measured by the Antonovsky Sense of Coherence Scale | Last day (i.e. expected 3rd or 4th day) of 5th cycle of chemotherapy after enrolment in study
  Self-report, registered once during 5th cycle of chemotherapy
Satisfaction with music intervention as measured by a Likert-type Scale (participants in music group only) | Last day (i.e. expected 3rd or 4th day) of 5th cycle of chemotherapy after enrolment in study
  Self-report, registered once during 5th cycle of chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Ilan Sanfi, PhD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Derived] Bradt J, Dileo C, Myers-Coffman K, Biondo J. Music interventions for improving psychological and physical outcomes in people with cancer. Cochrane Database Syst Rev. 2021 Oct 12;10(10):CD006911. doi: 10.1002/14651858.CD006911.pub4. PMID 34637527